CLINICAL TRIAL: NCT03131089
Title: Prospective Cohort Study for Development of Personalized Treatment Strategy Based on Biologic Tumor Behavior and Clinical Characteristics in Young Breast Cancer (YBC) Patients
Brief Title: Young Breast Cancer Cohort Study
Acronym: YBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Other Study IDs: 2013-04-005
Record Dates: First submitted 2017-04-16; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from breast cancer tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is prospective cohort study to investigate and identify comprehensively the clinicopathological features and long-term outcome of young breast cancer (YBC).

We have enrolled Breast cancer patients under 40 year-old and collected their baseline characteristics including tumor character, familiar history and other background information. Moreover, we have collected breast cancer tissue/blood sample for analyzing genetic characteristics, if patient agree to genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with breast cancer
2. Age under 40 year-old or diagnosis with breast cancer at pregnancy or within 1year after delivery
3. Obtained informed consent form

Exclusion Criteria:

1) Cannot understand or disagree to informed consent form

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Diagnosis with breast cancer
  2. Age under 40 year-old or diagnosis with breast cancer at pregnancy or within 1year after delivery
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-04-11 (Actual); Primary Completion 2018-02-17 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time to detect disease recurrence from surgery date

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No